CLINICAL TRIAL: NCT03459768
Title: Cohort Study on People Who Inject Drugs in Senegal
Acronym: CoDISEN
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: French National Agency for Research on AIDS and Viral Hepatitis (Other Government)
Responsible Party: Sponsor
Organization: ANRS, Emerging Infectious Diseases (Other Government)
Other Study IDs: ANRS 12334 CoDISEN
Record Dates: First submitted 2016-08-10; First posted 2018-03-09 (Actual); Last update posted 2021-06-08 (Actual); Status verified 2021-06

CONDITIONS: Drug Addiction; HIV/AIDS; Hepatitis C, Chronic; Hepatitis C, Acute; Hepatitis B, Chronic; Hepatitis B Acute; Tuberculosis; Sexually Transmitted Diseases; Psychiatric Disorder
MeSH Terms: conditions — Substance-Related Disorders; Acquired Immunodeficiency Syndrome; Hepatitis C, Chronic; Hepatitis C; Hepatitis B, Chronic; Tuberculosis; Sexually Transmitted Diseases; Mental Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — plasma and serum collected for biobank
Oversight: Data Monitoring Committee: No

SUMMARY:
The main purpose of the CoDISEN cohort study is to propose a model of prevention and care for HIV and viral hepatitis adapted to the needs of people who inject drugs (PWID) in Dakar, Senegal.

DETAILED DESCRIPTION:
THE UNODC estimated the number of consumers of injectable drugs at 1,02 millions in 2012 in Africa among which 12,1 % lived with HIV. Prevalences of HIV, chronic hepatitis C and B among people who inject drugs remain little documented in Sub-Saharan Africa. The transmission of HCV in Africa is mainly hospital-borne, bound to a precarious transfusional and therapeutic safety. However, the transmission by intravenous drug use emerges as a new stake in public health in urban areas. The report of a strong HIV prevalence in the population of PWID in the sub-region ( for example, In 2007, in the Cape Verde, prevalence of the HIV was 14 % in emprisoned PWID against 0,8 % in the general population) contributed to assert the reality of the use of intravenous drugs in the region and the vulnerability of this population. Senegal, a country with an concentrated HIV epidemic [0,5 % prevalence in 2012, WHO source] is the first country of western Africa to have measured prevalence of HIV (5,2 %), HBV (7,9 %) and HCV (23,3 %) in PWID (Study ANRS 12243). In view of these results, the Senegalese authorities introduced from October, 2011 in Dakar, activities of harm reduction by means of a mobile team of social workers and mediators allowing individual and collective activities of prevention, needle exchange program, references for care and follow-up, as well as a opioid substitution program in a methadone center (CEPIAD) located in Dakar, first of its kind in Western Africa. The objective of the present research project thus is to estimate the impact of a strategy of " test and treat " of HIV and harm reduction initiatives on the prevalence and incidence of HIV, HBV and HCV infections in an population of injectable drug consumers followed in the methadone center ( CEPIAD) of Dakar, Senegal

ELIGIBILITY:
Inclusion Criteria:

* being aged greater than or equal to 18 years or emancipated minor,
* Being or have been an injecting drug user and followed at the CEPIAD (methadone program)
* Living in the Dakar region for at least three months,
* Consenting to the study after individual information.

Exclusion Criteria:

* Mental impairment making it difficult or impossible to consent to the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Population of active injecting drug users who are seeking care at the CEPIAD, Dakar, Senegal.
Sampling Method: Non-Probability Sample
Enrollment: 208 (Actual)
Dates: Start 2016-08-24 (Actual); Primary Completion 2021-06-30 (Estimated); Study Completion 2021-06-30 (Estimated)

PRIMARY OUTCOMES:
incidence of HIV | 24 months
  number of participants infected with HIV at inclusion and acquiring HIV during follow-up

SECONDARY OUTCOMES:
incidence of hepatitis C infection (HCV) | 24 months
  number of participants infected with HCV at inclusion and acquiring HCV during follow-up
incidence of hepatitis B infection (HBV) | 24 months
  number of participants infected with HBV at inclusion and acquiring HBV during follow-up
incidence of relevant coinfections and comorbidities | 24 months
  number of patients developping sexually transmitted infections, tuberculosis and other conditions
  -% Test realized / test planned
Retention rate and its determinants | 24 months
  Number of participants retained in the cohort follow-up + analysis of determinants of retention
mortality rate and determinants | 24 months
  Number of participants dead during follow-up + analysis of determinants of death
  * evolution of CD4 and HIV viral load in participants with HIV and treated with ARVs, HBV viral load , and HCV viral load in participants with viral hepatitis B and C
  * Incidence of clinical events and biological of interest
Access to treatment of HCV, HBV infections and other coditions requiring specific therapeutical management | 24 months
  Number of patients treated for HIV, HBV, HCV and other medical conditions according to national or international guidelines recommendations
Effectiveness of tuberculosis regimens | 24 months
  Number of cured patients / number of patients initiating treatment

CONTACTS AND LOCATIONS:
Overall Officials: Pierre-Marie Girard, M.D., PhD, Principal Investigator — Inserm - Sorbonne Université; Moussa Seydi, M.D., Principal Investigator — CRCF - CHNU Fann
Locations (1):
- CEPIAD, Dakar, Senegal

IPD SHARING:
Plan to Share IPD: Yes
IPD that can be shared include study protocol, statistical analysis plan, inform consent form and anonymized database
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Duration of the study and 2 years after study closure
Access Criteria: Any sharing of information related to the study must be approved by the Scientific committee and the sponsor.